CLINICAL TRIAL: NCT01702480
Title: Effects of Medium-Chain Triglycerides on Cognitive Function in Older Subjects With Age-Related Cognitive Decline
Brief Title: Effects of Triglycerides on Age-Related Cognitive Function Decline in Older Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116713
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer's Disease
Keywords: Consumer Healthcare; Ketones; Medium Chain Triglycerides; Age related cognitive decline; GSK Nutrition
MeSH Terms: conditions — Alzheimer Disease; Ketosis | interventions — GSK2981710

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1: GSK2981710 10 gram (g) (Experimental): Eight subjects will receive single dose of GSK2981710 in the form of 10 g medium-chain triglycerides (MCT) powder daily for 14 days.
  Interventions: Drug: GSK2981710
- Part 1: GSK2981710 20 g (Experimental): Eight subjects will receive single dose of GSK2981710 in the form of 20 g MCT powder daily for 14 days.
  Interventions: Drug: GSK2981710
- Part 1: GSK2981710 30 g (Experimental): Eight subjects will receive single dose of GSK2981710 in the form of 30 g MCT powder daily for 14 days.
  Interventions: Drug: GSK2981710
- Part 1: GSK2981710 40 g (Experimental): Eight subjects will receive single dose of GSK2981710 in the form of 40 g MCT powder daily for 14 days.
  Interventions: Drug: GSK2981710
- Part 1: Placebo (Placebo Comparator): Eight subjects will receive single dose of matching placebo daily for 14 days.
  Interventions: Drug: Placebo
- Part 2: GSK2981710 (dose to be decided from Part 1) (Experimental): The subjects will receive single dose of GSK2981710 in the form of MCT powder (dose to be decided from Part 1) daily for 14 days.
  Interventions: Drug: GSK2981710
- Part 2: Placebo (Placebo Comparator): The subjects will receive single dose of matching placebo daily for 14 days..
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2981710 — Will be available as 10 g medium-chain triglycerides (MCT) powder sachet that will be mixed with 125 - 250 milliliters (ml) water in a shaker and taken within 15 minutes of completion of breakfast
  Arms: Part 1: GSK2981710 10 gram (g); Part 1: GSK2981710 20 g; Part 1: GSK2981710 30 g; Part 1: GSK2981710 40 g; Part 2: GSK2981710 (dose to be decided from Part 1)
Drug: Placebo — Will be available as matching powder that will be mixed with 125 - 250 milliliters (ml) water in a shaker and taken within 15 minutes of completion of breakfast
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
This is a single centre, 2 part study in older subjects. Part 1 (Pharmacokinetic [PK] Assessment) is a double blind, randomized, placebo-controlled 4-period crossover study investigating the PK profile of four different doses of GSK2981710. Eight subjects will receive a single dose of GSK2981710 10 gram (g), 20 g, 30 g, 40 g or placebo in the morning and have PK assessments (every 0.5 hrs up to 8 hrs post-dose) throughout the day in each period. Each subject will complete a total of four dosing sessions and 4 days of PK assessments in 2 weeks. The Part 1 PK data will be used for dose selection and pharmacodynamic (PD) assessment period in Part 2. If the data from Part 1 is inconclusive, an additional 8 subjects may be recruited and Part 1 repeated (possibly dropping some doses) to increase confidence. A subject's total participation in Part 1 of the study will last a maximum of approximately 7 weeks including screening. Subjects who have completed Part 1 may be screened for eligibility and enrolled for Part 2.

Part 2 (PD Assessment) is a double blind randomized, placebo-controlled 2-period crossover design with 14-day treatment periods investigating the efficacy (cognitive performance) and tolerability (gastrointestinal [GI] side effects) of single daily dose of GSK2981710 selected from Part 1. Part 2 of the study will include the Screening period, two Baseline assessments (6-8 days before each Treatment period) and two 14-day treatment periods separated by a minimum 7-day washout period and follow-up visit of 3 to 5 days. Approximately 50 to 80 subjects will be randomized to either GSK2981710 or placebo. The PD assessments will be performed on 6 occasions for each subject: at 2 baselines (6 to 8 days before Day 1 of each treatment period), post-dose on the Day 1 of each treatment period to assess acute effects and on Day 15 of each treatment period (which is the day after the final dose) to assess chronic effects. A subject's total participation in Part 2 of the study will last approximately up to 12 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals between the ages of 55 years and 80 years inclusive.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. Child-bearing potential and has a negative pregnancy test on each of the testing visits.
* Body weight >=50 kilogram (kg) in males and >=40 kg in females. Body mass index (BMI) in the range 18.0 to 29.9 kg/meter (m)^2.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Sufficiently fluent in English that they are able to understand written and spoken instructions in the opinion of the investigator.
* Supine blood pressure between 110/70 to 150/90 millimetres of mercury (mmHg) inclusive at screening. Patients with a current history of hypertension who are controlled on a stable regimen for at least 3 months prior to the study and are asymptomatic can be included.
* 12 lead electrocardiogram (ECG) without any clinically significant abnormality as judged by the Investigator, and QT interval corrected using Bazett's formula (QTcB) or QT interval corrected using Fridericia's formula (QTcF) <=450 millisecond (msec)
* Suitable for cannulation and with adequate venous access
* Aspartate aminotransferase (AST), Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* For Part 2: Performs below the cut-off level on the Wechsler logical memory test below the mean level of performance of young, healthy adults.
* For Part 2: Otherwise normal neuropsychological performance as indicated by performance above the required level on the MINI Mental State Examination (MMSE) (a score of 27 or above is eligible).

Exclusion Criteria:

* Previous or current medical condition, which as judged by the Investigator with consultation with the GSK Medical Monitor if required, may compromise subject safety or may interfere with the study procedures or the interpretation of data..
* Learning disability or learning disorder.
* Current history of Axis I psychiatric disorder as determined by MINI interview
* A drug dependence by the Diagnostic and Statistical Manual of Mental Disorders, Fourth (DSM-IV) criteria within the last 6 months as assessed by the Mini-international neuropsychiatric interview (MINI).
* A fall of at least 20 mm Hg systolic blood pressure within three minutes of standing upright at screening
* A positive pre-study human immunodeficiency virus (HIV), Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of alcohol or substance abuse or dependence in the 6 months prior to screening as determined by the investigator. Abuse of alcohol, defined for males, as an average weekly intake of greater than 21 units (or an average daily intake of greater than 3 units), or defined for females, as an average weekly intake of greater than 14 units (or an average daily intake of greater than 2 units). One unit is equivalent to a half-pint (220 milliliters [mL]) of beer or 1 (25 mL) measure of spirits or 1 glass (125 mL) of wine.
* Current smokers defined as regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Positive urine drug or alcohol breath test at screening or when tested at any of the study visits.
* Lactating females or pregnant females as determined by a positive urine/serum human chorionic gonadotropin (hCG) test at screening or when tested at any of the study visits.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the testing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Lactose intolerant or allergic to milk or soy products
* The subject is on a diet including any diet that restricts or modifies intake of a particular type of food, e.g. carbohydrates, proteins, fats, or is on a ketogenic diet.
* Fasting Triglycerides equal to or more than 4.5 millimoles per litre; (mmol/L) at screening
* Subject who, in the investigator/designee's judgement, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any evidence of suicidal ideation on any questionnaires e.g. type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) in the last 6 months.
* History of sensitivity or allergy to drug or components thereof, or other allergy, that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2012-11-05 (Actual); Primary Completion 2015-07-03 (Actual); Study Completion 2015-07-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Plasma BHB elevation time course of GSK2981710 | Baseline (Day 0 pre dose) and Day 1 post dose (per 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6, 6.5, 7, 7.5 and 8 hrs) of each of the 4 treatment periods.
  To select the dose of GSK2981710 that achieves the best PK profile, the duration of maximum elevation of beta-hydroxybutrate (BHB) will be measured.
Part 1: Area under the time concentration curve (AUC) of GSK2981710 | Baseline (Day 0 pre dose) and Day 1 post dose (per 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6, 6.5, 7, 7.5 and 8 hrs) of each of the 4 treatment periods.
  To select the dose of GSK2981710 that achieves the best PK profile the AUC of GSK2981710 will be measured.
Part 1: Maximum concentration (Cmax) of GSK2981710 | Baseline (Day 0 pre dose) and Day 1 post dose (per 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 5.5, 6, 6.5, 7, 7.5 and 8 hrs) of each of the 4 treatment periods.
  To select the dose of GSK2981710 that achieves the best PK profile the Cmax of GSK2981710 will be measured.
Part 2: Change from Baseline in performance on CANTAB Paired Associates Learning task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  To measure acute (after single dose) and chronic (after two weeks daily dosing) effects of GSK2981710 on cognition and neural function Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used. This test assesses visual memory and new learning
Part 2: Change from Baseline in performance on CANTAB Verbal Recognition Memory task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  To measure acute (after single dose) and chronic (after two weeks daily dosing) effects of GSK2981710 on cognition and neural function CANTAB will be used. This test assesses the participant's ability to recall as many of the words as possible immediately following the presentation of list of words.
Part 2: Change from Baseline in performance on CANTAB Spatial Working Memory (SWM) task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  To measure acute (after single dose) and chronic (after two weeks daily dosing) effects of GSK2981710 on cognition and neural function CANTAB will be used. This test assesses the participant's ability to retain spatial information and to manipulate remembered items in working memory.
Part 2: Change from Baseline in performance on CANTAB Rapid Visual Processing task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  To measure acute (after single dose) and chronic (after two weeks daily dosing) effects of GSK2981710 on cognition and neural function CANTAB will be used. This test assesses continuous performance and visual sustained attention.
Part 2: Change from Baseline in performance on CANTAB Reaction Time task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  To measure acute (after single dose) and chronic (after two weeks daily dosing) effects of GSK2981710 on cognition and neural function CANTAB will be used. This test measures of attention, and combines simple reaction time and choice reaction time elements
Part 2: Change from Baseline in performance on Source Memory Task | Baseline (Day 0) and Day 1 (post dose) and Day 15 (post dose) of both treatment periods.
  This test measures the participant's ability to recognize objects previously presented on a computer screen, and more importantly, to recall the spatial location of those objects.

SECONDARY OUTCOMES:
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by number of subjects with adverse events (AE)s | Part 1: 3 weeks; Part 2: 8 weeks
  Safety and tolerability parameters will include recording of AEs, in Part 1 and Part 2 of the study.
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by change from Baseline in ECG readings | Part 1: Baseline and 3 to 5 days post last dose in each of the 4 treatment periods.
  Safety and tolerability parameter will include the electrocardiogram (ECG) readings at Baseline (Day 0) and at end of Part 1 and Part 2 of the study. ECG will be performed at follow-up only if clinically indicated or pre-dose values are out of range as reviewed by the Principal Investigator or designee.
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by change from Baseline in laboratory values | Part 1: Baseline and 3 to 5 days post last dose in each of the 4 treatment periods.
  Safety and tolerability parameters will include laboratory (clinical chemistry, fasting blood glucose and hematological parameters) values at Baseline for Part 1 and Day 1 for Part 2 and at end of Part 1 and Part 2 of the study.
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by change from Baseline in vital signs | Part 1: Baseline and 3 to 5 days post last dose in each of the 4 treatment periods.
  Vital signs measurement include systolic and diastolic blood pressure, pulse rate and weight at Baseline (Part 2: Day 1) and at end of Part 1 and Part 2 of the study.
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by Gastrointestinal (GI) Symptom and stool diary | Part 1: Day -7 until Day 49.
  The subject will assess the GI symptom by capturing the information regarding GI symptoms, stool consistency and frequency in a self administered stool dairy card.
Part 1 and 2: Safety and tolerability of GSK2981710 as assessed by Liking Assessment | Part 1: Day 1 post dose of each of the 4 treatment periods.
  The subject used the liking assessment scale to assess the degree of liking for the GSK2981710.
Part 2: Change from Baseline in P300 EEG measurement | Baseline and Day 1 and Day 15 of each of the 2 treatment periods.
  The P300 (P3) is an electrophysiological index of neural processing that reflects a variety of cognitive processes elicited by a change in the sensory environment. Change from Baseline (Day 0) will be calculated as value at Day 1 and Day 15 minus the value at Day 0.
Part 2: Resting EEG measurement | Baseline and Day 1 and Day 15 of each of the 2 treatment periods.
  In this study the cognitive function will be assessed by measuring both high and low frequencies related to synchronized neuronal brain oscillations using resting electroencephalography (EEG).
Part 2: EEG measurement during Source Memory Task | Baseline and Day 1 and Day 15 of each of the 2 treatment periods.
  To measure the participant's ability to recognize objects previously presented on a computer screen, and more importantly, to recall the spatial location of those objects EEG will be used. The EEG is an electrophysiological measure of electrical neural activity.
Part 2: Correlation between systemic exposure of BHB and selected PD measurements | Day 1 and Day 15 of each of the 2 treatment periods.
  The correlation between systemic exposure (AUC, partial AUC) of BHB and selected PD measurements will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study 116713 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116713?search=study&b'study_ids=116713'#rs